CLINICAL TRIAL: NCT00748358
Title: An Open Label Phase II Study of Oral Treatment With Sunitinib (SUTENT) in Patients Suffering From Hormone Refractory Prostate Cancer After Progression With Docetaxel Based Regimen
Brief Title: An Open-label Phase II Study With SUTENT in Patients Suffering From Hormone Refractory Prostate Cancer
Acronym: PROSUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070404
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Prostatic Neoplasms; Neoplasms, Hormone-Dependent; Tumor Markers, Biological; Survival Rate; Disease-Free Survival
Keywords: metastatic prostate carcinoma; sunitinib [Substance Name]; Clinical Trial, Phase II [Publication Type]
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms, Hormone-Dependent | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug (Experimental): drug
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — 37.5 mg orally once daily, continuously, for 6 cycles of 6 consecutive weeks.Dose increase or reduction of 12.5 mg increments and change of schedule is recommended based on individual safety and tolerability.

SUMMARY:
as second-line treatment in metastatic prostate cancer, the present study will investigate the efficacy of sunitinib (SUTENT) given orally at a dose of 37.5 mg continuously, for 6 cycles of 6 consecutive weeks .Patients who are still responders after 6 cycles will be treated until disease progression, pain progression, unacceptable toxicity or death due to any cause.

Dose increase or reduction of 12.5 mg increments and change of schedule is recommended based on individual safety and tolerability.

Follow-up for up to 1 year from the last dose of sunitinib.

DETAILED DESCRIPTION:
* Antitumor efficacy of sunitinib will be assessed as follows:

  * PSA response rate and PSA progression according Working Group Criteria,
  * Variation of PSA doubling time (PSADT) before and after initiation of the treatment,
  * Objective response rate (ORR) according to RECIST criteria,
  * Clinical benefit,
  * Overall survival (OS).
* Pharmacokinetic endpoints will include sunitinib and its metabolite, SU012662, plasma levels and estimation of the population pharmacokinetic parameters as well as the inter-individual variability of these parameters, for a subgroup of 30 patients.
* The biological effects of sunitinib in patients with metastatic prostate carcinoma will be evaluated by measurements of the different biological markers that could be modulated by this antiangiogenic therapeutic, and could then predict and monitor disease progression and response to treatment:

  * Bone tumor markers: bone resorption markers (uCTX, uCTX, ICTP, CTX-MMP and TRACP-5b), bone formation markers (OC, PINP and BALP), osteoclastogenesis markers (OPG and RANKL) and parameters as calcium, phosphate, creatinine, albumin, PTH and 25(OH)D.
  * Angiogenesis markers: bFGF, SDF-1, VEGF-A, VEGFR1 and VEGFR2, CECs and CEPs, endothelial and platelet microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB/EC-approved informed consent
* Age 18 years or older
* Histologically confirmed prostate adenocarcinoma
* Metastatic HRPC
* Received prior castration by orchidectomy and/or LH-RH agonist with or without antiandrogen, antiandrogen withdrawal, monotherapy with estramustine, or other hormonal agents.
* Tumor disease must be progressive after a first line using docetaxel based chemotherapy, eventually in association with estramustine. Docetaxel based regimen may have been interrupted and restarted. Patient must have either measurable (RECIST criteria) or non-measurable (bone) disease and/or clinical progression (bone pain) and/or biological progression (PSA Working Group criteria).
* Discontinuation from previous chemotherapy and/or radiation therapy at least 4 weeks prior to treatment initiation
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Patient of child bearing potential must use effective contraception. Female partners of treated patients with child bearing potential must use oral contraceptives or intra uterine device (IUD)
* Life expectancy of at least 3 months
* Resolution of all acute toxic effects of any prior local treatment to NCI CTCAE grade 1
* Patients must have adequate organ functions defined
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patient covered by the National Health System

Exclusion Criteria:

* Prior treatment with sunitinib or other antiangiogenic agent
* More than 1 line of chemotherapy
* External beam radiotherapy for ≥ 50% of bone marrow
* Uncontrolled hypertension (systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg despite optimal medical management)
* Any of the following within 12 months prior to treatment initiation: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, thrombotic or embolic events such as cerebrovascular accident including transient ischemic attack
* Ongoing cardiac dysrhythmias of grade 2, atrial fibrillation of any grade
* Treatment with anticonvulsant agents and treatment with therapeutic doses of coumarin-derivative anticoagulants such as warfarin currently or within 2 weeks prior to first day of Sunitinib administration. Low dose of warfarin for deep vein thrombosis prophylaxis is permitted (up to 2 mg/day) and low molecular weight heparin is allowed
* Any medical condition that might interfere with oral medication absorption
* Known or suspected brain metastasis, or carcinomatous meningitis, or spinal cord compression
* Diagnosis of any second malignancy within the last 3 years, with the exception of treated basal cell or squamous cell carcinoma and pT1/a bladder cancer with no evidence of recurrent disease for 12 months
* Any acute or chronic medical or psychiatric disorder incompatible with the study
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness
* Treatment with others investigational drugs or participation in another clinical trial within the past 4 weeks, or concomitantly with this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) defined as the time from start of study treatment to first documentation of objective progressive disease, pain progression or to death on-study due to any cause. | 18 months

SECONDARY OUTCOMES:
Incidence and intensity of Adverse Events (NCI CTCAE version 3.0). | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: stephane OUDARD, professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service Oncologie Médicale, Hopital Europeen Georges Pompidou, Paris, France